CLINICAL TRIAL: NCT05702450
Title: A Randomized, Open, Parallel Phase I Clinical Study on the Comparison of Pharmacokinetics Characteristics of CM310 Recombinant Humanized Monoclonal Antibody Injection in Healthy Subjects
Brief Title: Study to Evaluate Pharmacokinetics, Safety and Efficacy of CM310
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM310-100002
Record Dates: First submitted 2023-01-12; First posted 2023-01-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P1 (Experimental): CM310, Subcutaneous
  Interventions: Biological: CM310
- Group P2 (Active Comparator): CM310, Subcutaneous, as the parallel control group
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — CM310 Recombinant Humanized Monoclonal Antibody Injection

SUMMARY:
This is a single-center, randomized, open study to evaluate the pharmacokinetics, safety and immunogenicity CM310 in healthy subjects.

DETAILED DESCRIPTION:
This study includes screening and treatment and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the study.
* Voluntarily participate in the study and sign the ICF.
* 18 years ≤ age ≤ 65 years, male and female.
* Willing to take effective contraceptive measures during the study period.

Exclusion Criteria:

* Plan to receive any major surgery during the study period.
* With malignant tumors within 5 years before screening.
* Positive results of alcohol breath test or urine drug abuse screening during screening period.
* Any reason that the investigator believes that will prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic: the maximum concentration (Cmax) | up to 57 days
  Concentration and exposure

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, Principal Investigator — Peking University Care Luzhong Hospital; Hong Wang, Principal Investigator — Peking University Care Luzhong Hospital
Locations (1):
- PKUCare Luzhong Hospital, Zibo, China